CLINICAL TRIAL: NCT03673605
Title: Efficacy and Safety of Rivaroxiban Compare With Vitamin K Antagonist Warfarin in Patients With Atrial Fibrillation and Mitral Stenosis Among Pakistani Population
Brief Title: Efficacy and Safety of Rivaroxiban Compare With Vitamin K Antagonist Warfarin
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients Enrollment
Sponsor: PharmEvo Pvt Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PE/NICVD/TS/Rivo/01
Record Dates: First submitted 2016-12-08; First posted 2018-09-17 (Actual); Last update posted 2018-09-17 (Actual); Status verified 2016-12

CONDITIONS: Mitral Valve Stenosis; Atrial Fibrillation
MeSH Terms: conditions — Mitral Valve Stenosis; Atrial Fibrillation | interventions — Rivaroxaban; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Rivaroxaban (Experimental)
  Interventions: Drug: Rivaroxaban 15 mg
- Warfarin (Active Comparator)
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Rivaroxaban 15 mg — Rivaroxiban in stroke prevention in patients with Mitral Stenosis and AF.
  Arms: Rivaroxaban
Drug: Warfarin — Warfarin in stroke prevention in patients with Mitral Stenosis and AF.
  Arms: Warfarin

SUMMARY:
Title: Efficacy and safety of rivaroxiban compare with vitamin K antagonist warfarin in patients with atrial fibrillation and mitral stenosis among Pakistani population.

DETAILED DESCRIPTION:
Atrial fibrillation is associated with an increase in the risk of ischemic stroke by a factor of four to five and accounts for up to 15% of strokes in persons of all ages and 30% in persons over the age of 80 years. The use of vitamin K antagonists is highly effective for stroke prevention in patients with non-valvular atrial fibrillation and is recommended for persons at increased risk. However, food and drug interactions necessitate frequent coagulation monitoring and dose adjustments, requirements that make it difficult for many patients to use such drugs in clinical practice.

Rivaroxaban is a direct factor Xa inhibitor that may provide more consistent and predictable anticoagulation than warfarin. It has been reported to prevent venous thromboembolism more effectively than enoxaparin in patients undergoing orthopedic surgery and was non-inferior to enoxaparin followed by warfarin in a study involving patients with established venous thrombosis. This trial was designed to compare once-daily oral rivaroxaban with dose-adjusted warfarin for the prevention of stroke and systemic embolism in patients with nonvalvular atrial fibrillation who were at moderate-to-high risk for stroke

ELIGIBILITY:
Inclusion Criteria:

* Both gender
* Age from 18 years up to 55 years
* Rheumatic MS (Mild moderate severe) Hemodynamic ally stable patients
* Associated AF or flutter documented on ECG
* Post PTMC or M com
* Not previously enrolled in any trial or study on NOACS
* Willing to participate

Exclusion Criteria:

* Rheumatic valve other than MS
* Prosthetic Mitral Valve Surgery
* Previous TIA or stroke
* Plan for valve replacement within six months
* Pregnancy
* History of bleeding complication
* High Risk of bleeding complication
* Allergic to study drug
* Anemia (HB less than 10 g/dl)
* Raised SGPT > 2xUNL
* Creatinine clearance <30ml/min
* Not willing to participate.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-30 (Actual); Primary Completion 2017-10-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Intracranial Bleeding and/or Recurrent Ischemic Lesion as Confirmed by MRI Imaging | 12 months
  Intracranial bleeding: symptomatic hemorrhage confirmed by CT or MRI or asymptomatic hemorrhage on follow-up GRE or SWI imaging at 1 month Recurrent ischemic lesion: symptomatic ischemic stroke confirmed by relevant neuroimagings or asymptomatic recurrent ischemic lesion on follow-up or FLAIR imaging at 12 month

SECONDARY OUTCOMES:
Adverse effects/complications of Rivaroxiban as compared to Warfarin in patients with Mitral Stenosis and AF. | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Cardiovascular, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes